CLINICAL TRIAL: NCT00193609
Title: A Phase II Trial of Oxaliplatin and Capecitabine in the Treatment of Patients With Relapsed/Refractory Carcinoma of Unknown Primary Site
Brief Title: Oxaliplatin and Capecitabine in the Treatment of Relapsed/Refractory Carcinoma of Unknown Primary Site
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Roche Pharma AG (Industry); Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI UNKPRI 14
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms, Unknown Primary
Keywords: Neoplasms, Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin/Capecitabine (Experimental): All patients received treatment with oxaliplatin 130mg/m2, given intravenously on day 1 of each 21 day cycle. Capecitabine 1000mg/m2 by mouth twice daily was administered on days 1-14 of each cycle.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m2 IV day 1 of 21 day cycle
  Other Names: Eloxatin
Drug: Capecitabine — 1000 mg/m2 by mouth twice daily on days 1-14 of each 21 day cycle
  Other Names: Xeloda

SUMMARY:
In this phase II trial, we will evaluate the feasibility and efficacy of the oxaliplatin/capecitabine combination in patients who have had one previous chemotherapy regimen for the treatment of carcinoma of unknown primary site. Patients who are relapsed after a previous response to treatment will be eligible, as well as those who were refractory to first-line therapy.

DETAILED DESCRIPTION:
All patients received treatment with oxaliplatin 130mg/m2, given intravenously on day 1 of each 21 day cycle. Capecitabine 1000mg/m2 PO BID was administered on days 1-14 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically confirmed carcinoma of unknown primary site
* Progressive disease after treatment with one previous chemotherapy regimen.
* Treatment with one previous immunotherapy or biotherapy regimen.
* No previous treatment with oxaliplatin, capecitabine, or 5-FU.
* Previous treatment with other platinum agents
* Patients must have measurable or evaluable disease
* ECOG Performance Status more than 2
* Adequate bone marrow, liver and kidney function
* Understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* History of treatment of any invasive malignancy within the last 5 years
* Coexistent medical illnesses
* Clinically significant cardiac disease
* Preexisting peripheral neuropathy > grade 1
* Lack of physical integrity of the upper gastrointestinal tract
* Pre-existing uncontrolled coagulopathy
* Women who are pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-09; Primary Completion 2008-04 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - AP&S Oncology & Hematology Northside, Terre Haute, Indiana
  - Greenview Regional Hospital, Bowling Green, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Oncology Hematology Care, Cincinnati, Ohio
  - Reading Hospital Regional Cancer Center, West Reading, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Burris HA 3rd, Shipley D, Farley C, Macias-Perez IM, Barton J, Greco FA. Oxaliplatin and capecitabine in the treatment of patients with recurrent or refractory carcinoma of unknown primary site: a phase 2 trial of the Sarah Cannon Oncology Research Consortium. Cancer. 2010 May 15;116(10):2448-54. doi: 10.1002/cncr.25029. PMID 20209610

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxaliplatin/Capecitabine
Started | 48
Completed | 44
Not Completed | 4
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention: All patients received treatment with oxaliplatin 130mg/m2, given intravenously on day 1 of each 21 day cycle. Capecitabine 1000mg/m2 by mouth twice daily was administered on days 1-14 of each cycle.
Arm/Group | Intervention
Number analyzed (Participants) | 48
Age Continuous [Median (Full Range); unit: years] | 59 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intervention
Number analyzed (Participants) | 44
months | 3.7 [2.6 to 9.7]

2. Secondary Outcome: Overall Survival
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until death.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intervention
Number analyzed (Participants) | 44
months | 9.7 [5.6 to 13.5]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 23/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=48)
vomiting (Gastrointestinal disorders) | 3 (3)
fever (General disorders) | 1 (1)
pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pancreatitis (Hepatobiliary disorders) | 1 (1)
pain (Gastrointestinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 4 (4)
disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper GI hemorrhage (Gastrointestinal disorders) | 1 (1)
left hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
adenocarcinoma of recturm (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
paralytic ileus (Gastrointestinal disorders) | 1 (1)
cardiopulmonary arrest (Cardiac disorders) | 1 (1)
CAD with ventricular tachycardia (Cardiac disorders) | 1 (1)
5-FU enteritis (Gastrointestinal disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
intrathecal catheter (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=48)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (20)
Anemia (Blood and lymphatic system disorders) | 14 (26)
Anorexia (Gastrointestinal disorders) | 19 (48)
Mood Alteration - Anxiety (Psychiatric disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (9)
Cold Sensitivity (General disorders) | 13 (23)
Constipation (Gastrointestinal disorders) | 14 (29)
Dehydration (Gastrointestinal disorders) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 25 (46)
Dizziness (Nervous system disorders) | 4 (7)
Edema - NOS (Blood and lymphatic system disorders) | 14 (39)
Fatigue (General disorders) | 34 (120)
Fever (General disorders) | 4 (4)
Hand-Foot (Skin and subcutaneous tissue disorders) | 8 (25)
Pain - Head (General disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Allergic Reaction (Immune system disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Infection - NOS (Infections and infestations) | 5 (7)
Mucositis/Stomatitis (Gastrointestinal disorders) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 35 (71)
Neuropathy (Nervous system disorders) | 25 (62)
Neutrophils (Blood and lymphatic system disorders) | 4 (12)
Pain (General disorders) | 16 (42)
Pulmonary - NOS (Respiratory, thoracic and mediastinal disorders) | 7 (14)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 8 (16)
Taste Alteration (Gastrointestinal disorders) | 4 (12)
Platelets (Blood and lymphatic system disorders) | 17 (59)
Vomiting (Gastrointestinal disorders) | 23 (39)
Weight Loss (Metabolism and nutrition disorders) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.